CLINICAL TRIAL: NCT05674097
Title: Blood Flow Path Reconstruction in Rectal Cancer After High IMA Ligation Through Preoperative and Postoperative Comparison by Manual Subtraction CTA
Brief Title: Blood Flow Path Reconstruction in Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Shandong First Medical University (Other)
Collaborators: Jinan Central Hospital (Other)
Responsible Party: Principal Investigator, Guoqin LIU, Director.Liu, Shandong First Medical University
Other Study IDs: 2020GQliu
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2022-12

CONDITIONS: Rectal Cancer; Surgery; Image
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
A total of 89 patients with distal sigmoid and rectal cancer were referred for observation and underwent MS-CTA between June 2020 and March 2022. The distribution of the left colic artery (LCA) was classified, and the presence of the accessory middle colic artery (AMCA) was assessed. Blood flow paths were planned preoperatively based on the classification of LCA branches. High ligation was performed during standard radical surgery. Intraoperatively, particular care was taken to preserve the bifurcation of the ascending and descending branches of the LCA. The planned blood flow paths were then compared with the actual postoperative blood flow paths to validate the previously proposed mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of distal sigmoid colon or rectal cancer
* cTNM stage confirmed as I-III on MRI or CT
* Undergoing laparoscopic anterior resection (LAR)

Exclusion Criteria:

* Arterial phase scanning initiated too early
* Unclear anatomic structure on imaging
* No postoperative enhanced CT

Ages: 39 Years to 81 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with distal sigmoid colon or rectal cancer and they were received routine laparoscopic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Six pattens of blood flow and AMCA based on the preoperative observation | 1 hour after the manual subtraction computed tomography angiography (MS-CTA) procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Guoqin LIU, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
It will be available when our paper is accepted.